CLINICAL TRIAL: NCT03171896
Title: Effect of the Involvement of a Medical Clown on the Labor Experience
Acronym: LaborClown
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: baruchPMC
Record Dates: First submitted 2016-10-25; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Affective Symptoms
MeSH Terms: conditions — Affective Symptoms | interventions — Laughter Therapy; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Medical clown
  Interventions: Other: clown
- No Intervention (Sham Comparator): No clown in the room
  Interventions: Other: Sham

INTERVENTIONS:
Other: clown — A medical clown will be offerred to the parturient and will spend time with her during labor as long as she will want it
  Arms: Intervention
Other: Sham — No clown will be present in the room during labor
  Arms: No Intervention

SUMMARY:
The experience of labor for a woman can be rewarding but can be traumatic. Medical clowning may alleviate the potential for trauma.

DETAILED DESCRIPTION:
The investigators plan to administer questionnaires to women who will agree to host a clown during their labor and to compare the feedback to those from women who did not.

ELIGIBILITY:
Inclusion Criteria:

Singleton pregnancy, Older than 18 years, Younger than 40 years, uncomplicated pregnancy

Exclusion Criteria:

Pregnancy complicated by PET, premature contractions Muktiple pregnancy, Older than 40 years, Younger than 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mood and satisfaction after labor | the day after delivery
  Women will answer questionairs which will be summarized and analyzed

IPD SHARING:
Plan to Share IPD: Yes
With the medical and general public